CLINICAL TRIAL: NCT00856986
Title: The Effect of Insulin Detemir in Combination With Liraglutide and Metformin Compared to Liraglutide and Metformin in Subjects With Type 2 Diabetes. A 26 Week, Randomised, Open-label, Parallel-group, Multicentre, Multinational Trial With a 26 Week Extension
Brief Title: The Effect of Insulin Detemir in Combination With Liraglutide and Metformin Compared to Liraglutide and Metformin in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1842; 2007-005317-19 (EudraCT Number)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2011-05-13 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Insulin Detemir; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lira 1.8 (Experimental): Subcutaneous administration of liraglutide 1.8 mg once daily in a forced 12 week run-in period + subject's own pre-trial metformin treatment at an unchanged dose and frequency (at least 1500 mg daily). Initial dose of liraglutide 0.6 mg/day with weekly increments of 0.6 mg until final dose of 1.8 mg/day was reached. Subjects were randomised to continue to receive liraglutide 1.8 mg once daily + metformin for 26 weeks plus 26 weeks extension, when the HbA1c assessment after run-in period was at least 7.0%
  Interventions: Drug: liraglutide; Drug: metformin
- Insulin detemir + Lira 1.8 (Experimental): Subcutaneous administration of liraglutide 1.8 mg once daily in a forced 12 week run-in period + subject's own pre-trial metformin treatment at an unchanged dose and frequency (at least 1500 mg daily). Initial dose of liraglutide 0.6 mg/day with weekly increments of 0.6 mg until final dose of 1.8 mg/day was reached. Subjects were randomised to continue to receive liraglutide 1.8 mg once daily + metformin in addition to individually adjusted insulin detemir for 26 weeks plus 26 weeks extension, when the HbA1c assessment after run-in period was at least 7.0%
  Interventions: Drug: liraglutide; Drug: insulin detemir; Drug: metformin
- Non-Randomised Lira 1.8 (Experimental): Subcutaneous administration of liraglutide 1.8 mg once daily in a forced 12 week run-in period + subject's own pre-trial metformin treatment at an unchanged dose and frequency (at least 1500 mg daily). Initial dose of liraglutide 0.6 mg/day with weekly increments of 0.6 mg until final dose of 1.8 mg/day was reached. Subjects continued to receive liraglutide 1.8 mg once daily + metformin for 26 weeks plus 26 weeks extension, when the HbA1c assessment after run-in period was below 7.0%
  Interventions: Drug: liraglutide; Drug: metformin
- Early Withdrawals Lira 1.8 (Other): Subcutaneous administration of liraglutide 1.8 mg once daily in a forced 12 week run-in period + subject's own pre-trial metformin treatment at an unchanged dose and frequency (at least 1500 mg daily). Initial dose of liraglutide 0.6 mg/day with weekly increments of 0.6 mg until final dose of 1.8 mg/day was reached. Due to withdrawals in the run-in period, subjects did not receive any further treatment in trial
  Interventions: Drug: liraglutide; Drug: metformin
- Intensified group (Other): Intensification of treatment with insulin detemir was offered at Weeks 26 and 38 for subjects with an HbA1c ≥ 8.0% in the randomised Lira 1.8 group and non-randomised liraglutide treatment group.
  Interventions: Drug: liraglutide; Drug: insulin detemir; Drug: metformin

INTERVENTIONS:
Drug: liraglutide — Liraglutide 1.8 mg/day for subcutaneous (under the skin) injection.
Drug: insulin detemir — Insulin detemir subcutaneous (under the skin) injection once daily. Dose will be titrated (individually adjusted) based on fasting self-measured plasma glucose levels according to a pre-specified algorithm
  Arms: Insulin detemir + Lira 1.8; Intensified group
Drug: metformin — Metformin tablets, at least 1500 mg/day

SUMMARY:
This trial is conducted in Europe and North America. The aim of this clinical trial is to assess and compare the effect of insulin detemir in combination with liraglutide and metformin versus liraglutide and metformin in subjects with type 2 diabetes. Subjects will continue their own pre-trial metformin treatment during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes, insulin naïve and treated with metformin as monotherapy for at least 3 months prior to screening, at a stable dose of at least 1500 mg/day or metformin (at least 1500 mg/day) and a sulfonylurea (less than or equal to half of the maximum approved dose), both at a stable dose for at least 3 months prior to screening. Previous short-term insulin treatment in connection with intercurrent illness is allowed at the discretion of the Investigator
* HbA1c 7.0-10.0% (both inclusive) for subjects on metformin monotherapy
* HbA1c 7.0-8.5% (both inclusive) for subjects on metformin in combination with a sulphonylurea

Exclusion Criteria:

* Previous treatment with insulin (except for short-term treatment in connection with intercurrent illness at the discretion of the Investigator)
* Treatment with glucose-lowering agent(s) other than stated in the inclusion criteria in a period of 3 months prior to screening
* Recurrent major hypoglycaemia or hypoglycaemic unawareness as judged by the Investigator
* Impaired kidney function
* Impaired liver function
* Uncontrolled treated/untreated hypertension
* Cancer or any clinically significant disease or disorder as judged by the Investigator
* Previous participation in the run-in phase of this trial. Re-screening is allowed once
* History of chronic pancreatitis or idiopathic pancreatitis

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (209):
- United States (52):
  - Novo Nordisk Investigational Site, Alexander City, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Los Gatos, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Jupiter, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Quincy, Illinois
  - Novo Nordisk Investigational Site, Chicago Heights, Indiana
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Methuen, Massachusetts
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Danville, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, State College, Pennsylvania
  - Novo Nordisk Investigational Site, Willkes Barre, Pennsylvania
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, Orem, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Belgium (2):
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Leuven
- Canada (7):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Ajax
- France (21):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Cahors
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Haguenau
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Perpignan
  - Novo Nordisk Investigational Site, Pessac
  - Novo Nordisk Investigational Site, Poitiers
  - Novo Nordisk Investigational Site, Reims
  - Novo Nordisk Investigational Site, Saint Quentin Cédex
  - Novo Nordisk Investigational Site, Saint-denis de La Reunion
  - Novo Nordisk Investigational Site, Saint-pierre de La Reunion
  - Novo Nordisk Investigational Site, Sète
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Tours
- Germany (34):
  - Novo Nordisk Investigational Site, Augsburg
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Bad Nauheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bremen
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Ebersheim
  - Novo Nordisk Investigational Site, Eisenach
  - Novo Nordisk Investigational Site, Erfurt
  - Novo Nordisk Investigational Site, Esslingen am Neckar
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Fulda
  - Novo Nordisk Investigational Site, Gifhorn
  - Novo Nordisk Investigational Site, Grevenbroich
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Jena
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Limburg
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Rosenheim
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Schkeuditz
  - Novo Nordisk Investigational Site, Sinsheim
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Wangen
- Italy (20):
  - Novo Nordisk Investigational Site, Ancona
  - Novo Nordisk Investigational Site, Caserta
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Catanzaro Lido
  - Novo Nordisk Investigational Site, Chiavari
  - Novo Nordisk Investigational Site, Cosenza
  - Novo Nordisk Investigational Site, Ferrara
  - Novo Nordisk Investigational Site, Lanciano
  - Novo Nordisk Investigational Site, Matera (mt)
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Monserrato, Cagliari
  - Novo Nordisk Investigational Site, Monza
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Piacenza
  - Novo Nordisk Investigational Site, Primo Piano Palazzina Ambulato
  - Novo Nordisk Investigational Site, Ravenna
  - Novo Nordisk Investigational Site, Reggio Calabria
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Terni
  - Novo Nordisk Investigational Site, Treviglio
- Netherlands (19):
  - Novo Nordisk Investigational Site, Amersfoort
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Beek
  - Novo Nordisk Investigational Site, Delft
  - Novo Nordisk Investigational Site, Doetinchem
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Heerlen
  - Novo Nordisk Investigational Site, Hoofddorp
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Leiden
  - Novo Nordisk Investigational Site, Leiderdorp
  - Novo Nordisk Investigational Site, Lichtenvoorde
  - Novo Nordisk Investigational Site, Lieshout
  - Novo Nordisk Investigational Site, Oude Pekela
  - Novo Nordisk Investigational Site, Utrecht
  - Novo Nordisk Investigational Site, Voorburg
  - Novo Nordisk Investigational Site, Wildervank
  - Novo Nordisk Investigational Site, Winschoten
- Puerto Rico (3):
  - Novo Nordisk Investigational Site, Bayamón
  - Novo Nordisk Investigational Site, Carolina
  - Novo Nordisk Investigational Site, Trujillo Alto
- Spain (23):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Badajoz
  - Novo Nordisk Investigational Site, Badalona
  - Novo Nordisk Investigational Site, Bilbao
  - Novo Nordisk Investigational Site, Cadiz
  - Novo Nordisk Investigational Site, Cartagena
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Girona
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Majadahonda
  - Novo Nordisk Investigational Site, Pamplona
  - Novo Nordisk Investigational Site, Pontevedra
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, Salamanca
  - Novo Nordisk Investigational Site, San Juan
  - Novo Nordisk Investigational Site, San Sebastián de los Reyes
  - Novo Nordisk Investigational Site, Santa Cruz de Tenerife
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Tarrasa
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Xátiva
  - Novo Nordisk Investigational Site, Zaragoza
- United Kingdom (28):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Ashton-under-Lyne
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Derby
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Inverness
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Londonderry
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Nuneaton
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Rugby
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Welwyn Garden City

REFERENCES:
- [Result] DeVries JH, Bain SC, Rodbard HW, Seufert J, D'Alessio D, Thomsen AB, Zychma M, Rosenstock J; Liraglutide-Detemir Study Group. Sequential intensification of metformin treatment in type 2 diabetes with liraglutide followed by randomized addition of basal insulin prompted by A1C targets. Diabetes Care. 2012 Jul;35(7):1446-54. doi: 10.2337/dc11-1928. Epub 2012 May 14. PMID 22584132
- [Result] Rosenstock J, Rodbard HW, Bain SC, D'Alessio D, Seufert J, Thomsen AB, Svendsen CB, DeVries JH; Liraglutide-Detemir Study Group. One-year sustained glycemic control and weight reduction in type 2 diabetes after addition of liraglutide to metformin followed by insulin detemir according to HbA1c target. J Diabetes Complications. 2013 Sep-Oct;27(5):492-500. doi: 10.1016/j.jdiacomp.2013.04.008. Epub 2013 Jun 6. PMID 23746555
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 202 centres in 9 countries: Belgium (2), Canada (7), France (19), Germany (37), Italy (18), the Netherlands (16), Spain (14), the United Kingdom (32) and the United States (57)
Pre-assignment Details: Subjects on metformin and/or sulpholynurea treatment underwent a 12-week run-in period with liraglutide + metformin. Subjects not achieving an HbA1c below 7% were randomised to liraglutide + metformin treatment with/without insulin detemir. Subjects achieving an HbA1c below 7% continued liraglutide + metformin treatment.
Period: Run-in Period, Weeks -12-0
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Started | 161 | 162 | 498 | 167 | 0
Completed | 161 | 162 | 498 | 0 (Subjects who withdrew during run-in and before randomisation were Early Withdrawals) | 0
Not Completed | 0 | 0 | 0 | 167 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 92 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 24 | 0
Not completed — Withdrawal Criteria | 0 | 0 | 0 | 10 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 11 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 6 | 0
Not completed — Unclassified | 0 | 0 | 0 | 24 | 0
Period: Main Period, Weeks 0-26
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Started | 161 | 162 | 498 | 0 | 0
Completed | 127 | 144 | 470 | 0 | 0
Not Completed | 34 | 18 | 28 | 0 | 0
Not completed — Adverse Event | 6 | 4 | 9 | 0 | 0
Not completed — Protocol Violation | 4 | 5 | 7 | 0 | 0
Not completed — Withdrawal Criteria | 11 | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0 | 0
Not completed — Lack of Efficacy | 5 | 2 | 0 | 0 | 0
Not completed — Unclassified | 7 | 6 | 7 | 0 | 0
Period: Extension Period, Weeks 26-52
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Started | 127 (Subjects with HbA1c ≥8.0% who accepted intensification with detemir = 17 (Intensified Group)) | 144 | 470 (Subjects with HbA1c ≥8.0% who accepted intensification with detemir = 7 (Intensified Group)) | 0 | 0
Enrolled in Extension | 122 | 140 | 461 | 0 | 0
Completed | 108 | 130 | 432 | 0 | 0
Not Completed | 19 | 14 | 38 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 10 | 0 | 0
Not completed — Protocol Violation | 6 | 2 | 5 | 0 | 0
Not completed — Withdrawal Criteria | 2 | 0 | 8 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 2 | 0 | 0
Not completed — Lack of Efficacy | 4 | 2 | 2 | 0 | 0
Not completed — Unclassified | 4 | 2 | 11 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group | Total
Number analyzed (Participants) | 161 | 162 | 498 | 166 | 24 | 1011
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.8) | 57 (9.5) | 56.7 (9.7) | 58.7 (10.8) | 54.3 (10.3) | 56.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 74 | 216 | 75 | 11 | 448
  Male | 89 | 88 | 282 | 91 | 13 | 563
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 48 | 28 | 5 | 128
  Not Hispanic or Latino | 136 | 140 | 450 | 138 | 19 | 883
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 4 | 5 | 4 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 17 | 8 | 19 | 11 | 1 | 56
  White | 141 | 144 | 470 | 146 | 22 | 923
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 4 | 5 | 1 | 16
Height [Mean (Standard Deviation); unit: meter] | 1.7 (0.1) | 1.69 (0.11) | 1.7 (0.1) | 1.68 (0.1) | 1.72 (0.09) | 1.69 (0.1)
Body weight [Mean (Standard Deviation); unit: kg] — At Week -12
  kg | 98.6 (21.3) | 99.5 (21.2) | 99 (20.8) | 90.2 (18.5) | 109 (25.7) | 99 (21)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — At Week -12
  kg/m^2 | 33.9 (6) | 34.9 (6.3) | 34.4 (6.7) | 31.8 (6) | 36.5 (7.7) | 34.4 (6.5)
Diabetes History [Mean (Standard Deviation); unit: years] | 8.5 (6) | 8.6 (5.8) | 6.6 (5.7) | 8.4 (6.4) | 6.8 (5.4) | 7.4 (5.8)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage point of total HbA1c] — At Week -12
  Percentage point of total HbA1c | 8.3 (0.8) | 8.2 (0.7) | 7.7 (0.7) | 8 (0.8) | 8.4 (0.7) | 7.9 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — At Week -12
  mmol/L | 10.3 (2.5) | 10.2 (2.4) | 9.2 (1.8) | 9.5 (3) | 10.4 (2.3) | 9.6 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Randomisation in Glycosylated Haemoglobin A1c (HbA1c) at Week 26.
Time Frame: Week 0 (Randomisation), week 26
Population: The FAS (Full Analysis Set) using LOCF (Last Observation Carried Forward) is all randomised subjects with at least one of any efficacy value after the randomisation visit (baseline)
Measure: Least Squares Mean (Standard Error); unit: Percentage point of total HbA1c
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 149 | 160 | 0 | 0 | 0
Percentage point of total HbA1c | 0.02 (0.07) | -0.51 (0.07) |  |  |
Statistical Analysis 1: Comparison: Lira 1.8 vs Insulin Detemir + Lira 1.8; The estimated treatment difference between Detemir+Lira 1.8 and Lira 1.8 as well as 95% confidence interval and p-value were calculated by an ANCOVA model with treatment, country and previous OAD as fixed factors and baseline value as covariate. The p-value reflects a two-sided test for the null hypothesis of no difference between the two treatment groups with a significance level of 5% and with the power of 90%; Test type: Superiority or Other; ANCOVA; Estimated Treatment Difference, LSMean = -0.52, 95% CI [-0.68 to -0.36]

2. Secondary Outcome: Mean Change From Randomisation in Glycosylated Haemoglobin A1c (HbA1c) at Week 52 (for Intensified Subjects in Original Treatment Group)
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage point of total HbA1c
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 149 | 160 | 0 | 0 | 0
Percentage point of total HbA1c | -0.1 (0.09) | -0.51 (0.09) |  |  |
Statistical Analysis 1: Comparison: Lira 1.8 vs Insulin Detemir + Lira 1.8; The estimated treatment difference between Detemir+Lira 1.8 and Lira 1.8 as well as 95% confidence interval and p-value were calculated by an ANCOVA model with treatment, country and previous OAD as fixed factors and baseline value as covariate. The p-value reflects a two-sided test for the null hypothesis of no difference between the two treatment groups with a significance level of 5%; Test type: Superiority or Other; ANCOVA; Estimated Treatment Difference, LSMean = -0.41, 95% CI [-0.6 to -0.21] — The analysis values for intensified Lira 1.8 mg subjects were kept in the treatment group and the last observation carried forward (LOCF) method was applied

3. Secondary Outcome: Mean Change From Randomisation in Glycosylated Haemoglobin A1c (HbA1c) at Week 52 (Values Before Intensification as LOCF)
Time Frame: Week 0, Week 52
Population: The FAS (Full Analysis Set) includes LOCF of last observation before intensification for randomised Lira 1.8 mg treatment group subjects who were intensified.
Measure: Least Squares Mean (Standard Error); unit: Percentage point of total HbA1c
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 149 | 160 | 0 | 0 | 0
Percentage point of total HbA1c | 0.01 (0.09) | -0.5 (0.09) |  |  |
Statistical Analysis 1: Comparison: Lira 1.8 vs Insulin Detemir + Lira 1.8; Test type: Superiority or Other; ANCOVA; Estimated treatment difference, LS mean = -0.51, 95% CI [-0.7 to -0.31] — The mean change in HbA1c from randomisation to week 52 was analysed including the values before intensification as LOCF for intensified subjects

4. Secondary Outcome: Mean Change From Randomisation in Fasting Plasma Glucose at Week 26
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 154 | 160 | 0 | 0 | 0
mmol/L | -0.39 (0.19) | -2.12 (0.19) |  |  |

5. Secondary Outcome: Mean Change From Randomisation in Fasting Plasma Glucose at Week 52
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 154 | 160 | 0 | 0 | 0
mmol/L | -0.14 (0.21) | -1.91 (0.21) |  |  |

6. Secondary Outcome: Mean Change From Randomisation in 7-point Plasma Glucose Profile (Self-measured) at Week 26
Description: Calculated as an estimate of the change in mean prandial increment of plasma glucose after breakfast, lunch and dinner (from baseline/randomisation (week 0) to 26 weeks), respectively. Prandial increments of plasma glucose were calculated as the difference between glucose values measured before and after each of these three meals, respectively.
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 133 | 144 | 0 | 0 | 0
mmol/L
  Change at Breakfast, N=133, 144 | -0.97 (0.26) | -2.09 (0.26) |  |  |
  Change at Lunch, N= 134, 143 | -0.83 (0.22) | -1.43 (0.22) |  |  |
  Change at Dinner, N= 133, 139 | -0.48 (0.24) | -1.18 (0.24) |  |  |

7. Secondary Outcome: Mean Change From Randomisation in 7-point Plasma Glucose Profile (Self-measured) at Week 52
Description: Calculated as an estimate of the change in mean prandial increment of plasma glucose after breakfast, lunch and dinner (from baseline (week 0) to 52 weeks), respectively. Prandial increments of plasma glucose were calculated as the difference between glucose values measured before and after each of these three meals, respectively.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 136 | 148 | 0 | 0 | 0
mmol/L
  Change at Breakfast, N=148, 135 | -0.68 (0.25) | -2.43 (0.25) |  |  |
  Change at Lunch, N= 145, 136 | -0.51 (0.25) | -1.14 (0.25) |  |  |
  Change at Dinner, N= 144, 135 | -0.96 (0.26) | -1.4 (0.25) |  |  |

8. Secondary Outcome: Mean Change From Randomisation in Fasting Insulin at Week 26
Time Frame: Week 0 (Randomisation), Week 26
Population: Data on fasting insulin could not be obtained for the insulin detemir+liraglutide 1.8 mg+metformin (Detemir + Lira 1.8 group) treated subjects due to cross-reactivity between insulin detemir and the insulin assay. Data from both goups were therefore not further investigated by ANCOVA why no data is presented for this endpoint.
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Mean Change From Randomisation in Fasting Insulin at Week 52
Time Frame: Week 0 (Randomisation), Week 52
Population: as for outcome 8
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Mean Change From Randomisation in Fasting Pro-insulin at Week 26.
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 135 | 152 | 0 | 0 | 0
pmol/L | -1.12 (3.27) | -9.78 (3.22) |  |  |

11. Secondary Outcome: Mean Change From Randomisation in Fasting Pro-insulin at Week 52
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 139 | 152 | 0 | 0 | 0
pmol/L | 1.47 (3.08) | -4 (3.08) |  |  |

12. Secondary Outcome: Mean Change From Randomisation in Fasting C-peptide at Week 26.
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 136 | 149 | 0 | 0 | 0
mmol/L | -0.08 (0.04) | -0.32 (0.04) |  |  |

13. Secondary Outcome: Mean Change From Randomisation in Fasting C-peptide at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 139 | 150 | 0 | 0 | 0
mmol/L | 0.02 (0.05) | -0.34 (0.05) |  |  |

14. Secondary Outcome: Mean Changes From Randomisation in Cholesterol Lipids at Week 26.
Description: Cholesterol Lipids cover: Total Cholesterol, Low-density Lipoprotein Cholesterol (LDL-C), Very Low Density Lipoprotein Cholesterol (VLDL-C), High Density Lipoprotein Cholesterol (HDL-C)
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 141 | 152 | 0 | 0 | 0
mmol/L
  Change in Total Cholesterol | 0.04 (0.07) | 0.05 (0.07) |  |  |
  Change in LDL-C | -0.04 (0.06) | -0.03 (0.06) |  |  |
  Change in VLDL-C | 0.05 (0.03) | 0.01 (0.03) |  |  |
  Change in HDL-C | 0.02 (0.01) | 0.05 (0.01) |  |  |

15. Secondary Outcome: Mean Changes From Randomisation in Cholesterol Lipids at Week 52.
Description: as for outcome 14
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 141 | 153 | 0 | 0 | 0
mmol/L
  Change in Total Cholesterol | -0.02 (0.08) | -0.03 (0.08) |  |  |
  Change in LDL-C | -0.08 (0.07) | -0.1 (0.07) |  |  |
  Change in VLDL-C | 0.03 (0.04) | -0.03 (0.04) |  |  |
  Change in HDL-C | 0.02 (0.02) | 0.07 (0.02) |  |  |

16. Secondary Outcome: Mean Change From Randomisation in Lipids: Triglycerides at Week 26
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 141 | 151 | 0 | 0 | 0
mmol/L | -0.24 (0.11) | -0.33 (0.11) |  |  |

17. Secondary Outcome: Mean Change From Randomisation in Lipids: Triglycerides at Week 52
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 141 | 152 | 0 | 0 | 0
mmol/L | -0.22 (0.11) | -0.37 (0.11) |  |  |

18. Secondary Outcome: Mean Change From Randomisation in Lipids: Free Fatty Acids (FFA) at Week 26
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 131 | 140 | 0 | 0 | 0
mmol/L | -0.03 (0.02) | -0.11 (0.02) |  |  |

19. Secondary Outcome: Mean Change From Randomisation in Lipids: Free Fatty Acids (FFA) at Week 52
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 133 | 141 | 0 | 0 | 0
mmol/L | -0.03 (0.03) | -0.07 (0.03) |  |  |

20. Secondary Outcome: Mean Change From Randomisation in Body Weight at Week 26
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 157 | 162 | 0 | 0 | 0
kg | -0.95 (0.31) | -0.16 (0.31) |  |  |

21. Secondary Outcome: Mean Change From Randomisation in Body Weight at Week 52
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 157 | 162 | 0 | 0 | 0
kg | -1.02 (0.41) | -0.05 (0.42) |  |  |

22. Secondary Outcome: Mean Change From Randomisation in Waist Circumference at Week 26.
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 148 | 160 | 0 | 0 | 0
cm | -0.66 (0.46) | -0.78 (0.46) |  |  |

23. Secondary Outcome: Mean Change From Randomisation in Waist Circumference at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: participants
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 148 | 160 | 0 | 0 | 0
participants | -0.83 (0.54) | -0.83 (0.53) |  |  |

24. Secondary Outcome: Mean Change From Randomisation in Hip Circumference at Week 26
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 148 | 160 | 0 | 0 | 0
cm | -0.36 (0.46) | -0.38 (0.45) |  |  |

25. Secondary Outcome: Mean Change From Randomisation in Hip Circumference at Week 52
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 148 | 160 | 0 | 0 | 0
cm | -0.79 (0.5) | -0.28 (0.49) |  |  |

26. Secondary Outcome: Mean Change From Randomisation in Waist to Hip Ratio at Week 26
Description: Waist to Hip Ratio is calculated by dividing Waist circumference with Hip circumference
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm/cm
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 148 | 160 | 0 | 0 | 0
cm/cm | -0.00356 (0.004071) | -0.00332 (0.004032) |  |  |

27. Secondary Outcome: Mean Change From Randomisation in Waist to Hip Ratio at Week 52
Description: Waist to Hip Ratio is calculated by dividing Waist circumference with Hip circumference
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm/cm
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 148 | 160 | 0 | 0 | 0
cm/cm | -0.00146 (0.004165) | -0.00438 (0.004126) |  |  |

28. Secondary Outcome: Mean Change From Randomisation in Blood Pressure (Systolic and Diastolic) at Week 26.
Time Frame: Week 0 (Randomisation), Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 157 | 162 | 0 | 0 | 0
mmHg
  Systolic Blood Pressure | 1.11 (1.22) | 0.41 (1.23) |  |  |
  Diastolic Blood Pressure | -1.1 (0.77) | -0.4 (0.78) |  |  |

29. Secondary Outcome: Mean Change From Randomisation in Blood Pressure (Systolic and Diastolic) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 157 | 162 | 0 | 0 | 0
mmHg
  Systolic Blood Pressure | -0.74 (1.2) | 0.16 (1.21) |  |  |
  Diastolic Blood Pressure | -0.66 (0.78) | 0.11 (0.79) |  |  |

30. Secondary Outcome: Adverse Events From Run-in (Week -12) to Week 52
Time Frame: Run-in (week -12) to Week 52
Population: The Safety Analysis Set included all exposed subjects
Measure: Number; unit: events
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 159 | 163 | 499 | 166 | 24
events | 716 | 845 | 2389 | 383 | 30

31. Secondary Outcome: Hypoglycaemic Episodes (Excluding Outlier Subject), Weeks 0-26
Description: Number of hypoglycaemic episodes from Week 0 to Week 26, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: weeks 0-26
Population: The Safety Analysis Set included all exposed subjects. An outlier subject from the lira 1.8 group, who experienced an extreme number of minor and symptoms only hypoglycaemic episodes was excluded from this analysis.
Measure: Number; unit: episodes
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 158 | 163 | 499 | 0 | 0
episodes
  Major | 0 | 0 | 0 |  |
  Minor | 2 | 22 | 31 |  |
  Symptoms only | 9 | 19 | 26 |  |

32. Secondary Outcome: Hypoglycaemic Episodes Weeks 0-52
Description: Number of hypoglycaemic episodes from Week 0 to Week 52, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Week 0-52
Population: as for outcome 31
Measure: Number; unit: episodes
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Number analyzed (Participants) | 159 | 163 | 499 | 0 | 24
episodes
  Major | 0 | 0 | 0 |  | 0
  Minor | 4 | 33 | 53 |  | 1
  Symptoms only | 14 | 57 | 42 |  | 2
  Unknown | 0 | 1 | 2 |  | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 64 weeks (from run-in to week 52).
Description: The Safety Analysis Set included all exposed subjects
Arm/Group | Lira 1.8 | Insulin Detemir + Lira 1.8 | Non-Randomised Lira 1.8 | Early Withdrawals Lira 1.8 | Intensified Group
Serious Adverse Events (participants affected / at risk) | 11/159 | 17/163 | 62/499 | 6/166 | 1/24
Other Adverse Events (participants affected / at risk) | 100/159 | 102/163 | 310/499 | 122/166 | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lira 1.8 (N=159) | Insulin Detemir + Lira 1.8 (N=163) | Non-Randomised Lira 1.8 (N=499) | Early Withdrawals Lira 1.8 (N=166) | Intensified Group (N=24)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter Gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interverterbal Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Interverterbal Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign Intracranial Hypertension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Macular Ischaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular Oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Squamous Cell Carcinoma Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor Peripheral Circulation (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid ccell hyperplasia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECG abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECG change (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.8 (N=159) | Insulin Detemir + Lira 1.8 (N=163) | Non-Randomised Lira 1.8 (N=499) | Early Withdrawals Lira 1.8 (N=166) | Intensified Group (N=24)
Nasopharyngitis (Infections and infestations) | 40 (57) | 33 (45) | 72 (97) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 26 (29) | 29 (42) | 74 (108) | 21 (25) | 1 (1)
Nausea (Gastrointestinal disorders) | 37 (51) | 30 (40) | 136 (204) | 66 (72) | 1 (1)
Lipase Increased (Investigations) | 16 (17) | 26 (27) | 55 (60) | 6 (7) | 4 (4)
Headache (Nervous system disorders) | 23 (41) | 21 (54) | 73 (144) | 13 (22) | 2 (2)
Vomiting (Gastrointestinal disorders) | 19 (21) | 17 (26) | 50 (113) | 21 (25) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 8 (11) | 10 (11) | 42 (54) | 33 (42) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (11) | 8 (10) | 25 (30) | 11 (11) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 8 (11) | 6 (7) | 14 (17) | 5 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (14) | 13 (13) | 21 (24) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (10) | 12 (13) | 15 (16) | 6 (8) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (6) | 26 (30) | 4 (5) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (5) | 17 (19) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 9 (9) | 13 (13) | 50 (53) | 17 (17) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right not to release data until specified milestones, e.g. a clinical trial report is available. This includes the right not to release interim results from clinical trials.

At the end of the trial, one or more manuscripts for publication will be prepared in collaboration between Investigator(s) and Novo Nordisk. Novo Nordisk will not suppress or veto publications. Novo Nordisk reserves the right to postpone publication for a short time to protect intellectual property.